CLINICAL TRIAL: NCT01532284
Title: The Eshre Study Into The Evaluation of Oocyte Euploidy by Microarray Analysis
Acronym: ESTEEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Society of Human Reproduction and Embryology (Other)
Responsible Party: Principal Investigator, Karen Sermon, Prof. dr., European Society of Human Reproduction and Embryology
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Screening
Other Study IDs: ESHRE-ESTEEM
Record Dates: First submitted 2012-02-07; First posted 2012-02-14 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Aneuploid Oocytes
Keywords: aneuploid oocytes; ICSI; IVF; Polar Body Biopsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polar Body Biopsy (Experimental): PB biopsy (PBB) will be performed between 9 and 12 hours after ICSI using laser or the mechanical procedure. PB1 and PB2 will be removed simultaneously (both at the same time) and transferred to different tubes for the chromosomal analysis.
  Interventions: Other: Polar Body Biopsy
- No Polar Body Biopsy (No Intervention)

INTERVENTIONS:
Other: Polar Body Biopsy — PB biopsy (PBB) will be performed between 9 and 12 hours after ICSI using laser or the mechanical procedure. PB1 and PB2 will be removed simultaneously (both at the same time) and transferred to different tubes for the chromosomal analysis.
  Arms: Polar Body Biopsy

SUMMARY:
A pragmatic, multicentre, randomized double-blind controlled trial with an intention-to-treat analysis, of the use of preimplantation genetic screening (PGS) for aneuploidy by means of microarray comparative genomic hybridization (CGH) for the chromosomal analysis of the polar bodies (PB) of oocytes collected after ovarian stimulation for in vitro fertilization (IVF), and with the intention to assess the genetic competence of oocytes of advanced biological age, and the effect of this technique on reproductive outcome.

ELIGIBILITY:
Inclusion Criteria:

* infertility as an indication for IVF or ICSI;
* patients between their 36th and 41st birthdays (at time of signing ICF i.e. max 40years and 364days at the day of signing the informed consent);
* BMI range 18 to 30 kgs per m2;
* patients prepared to accept transfer of up to two embryos;
* absence of any type of genetic abnormality in the patient's personal and family history;
* normal karyotype (optional)

Exclusion Criteria:

* treatment involving donor oocytes (donor sperm is allowed subject to local practice and regulations and provided karyotype of the sperm donor is available and normal);
* menstrual irregularity (<24 and >35 days);
* three or more previous failed IVF or ICSI cycles, with the present partner. (Definition of a failed cycle: 'absence of a clinical pregnancy relating to a treatment with embryo transfer resulting from oocyte retrieval for the current intended pregnancy and with the current partner; the transfers include transfers of fresh and frozen within this treatment; clinical pregnancy is defined as the presence of a gestational sac at the earliest ultrasound and includes early clinical miscarriage, late miscarriage and clinically confirmed extrauterine pregnancy, and excludes preclinical miscarriage (biochemical pregnancy); -
* three or more clinical miscarriages;
* poor response in any previous cycle;
* low ovarian reserve (At least one of the following two features must be present: (1) a previous poor ovarian response (≤ 3 oocytes with a conventional stimulation 119 protocol); (2) an abnormal ovarian reserve test (i.e. AFC < 5 follicles or AMH < 0,5 ng/mL)* (adapted from Ferraretti et al., 2011);
* cycles requiring surgical sperm recovery procedures;
* total asthenozoospermia and/or globozoospermia.
* any type of genetic abnormality or family history of genetic abnormality in subject or partner

Ages: 36 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 396 (Actual)
Dates: Start 2012-02; Primary Completion 2016-12 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
To improve live birth rates. | up to 1 year after birth
  This trial has two primary aims among women with advanced maternal age (1) to improve live birth rates and (2) to assess the prediction value of having no euploid oocytes in future ART cycles.
To assess the prediction value of having no euploid oocytes in future ART cycles. | Up to 1 year after birth
  This trial has two primary aims among women with advanced maternal age (1) to improve live birth rates and (2) to assess the prediction value of having no euploid oocytes in future ART cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sermon, Prof. dr., Principal Investigator — ESHRE
Locations (8):
- Centre for Reproductive Medicine BRUSSELSIVF and Centre Medical Genetics, Vrije Universiteit Brussel, Brussels, Belgium
- Germany (3):
  - Department of Gynecological Endocrinology and Reproductive Medicine, University of Bonn, Bonn, Germany, Bonn
  - gyn-medicum Göttingen; Zentrum für Kinderwunsch, Göttingen
  - UNIVERSITÄTSKLINIKUM Schleswig-Holstein - Sektion für gynäkologische Endokrinologie und Reproduktionsmedizin, Lübeck
- Department of Medical Genetics, Athens University/Genesis Athens Clinic, Greece, Athens, Greece
- Medical Genetics Institute, Shaare Zedek Medical Center and IVF Unit, Jerusalem, Israel
- Department of Reproductive Medicine, S.I.S.Me.R., Reproductive Medicine Unit,, Bologna, Italy
- Institut Universitari Dexeus, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Verdyck P, Altarescu G, Santos-Ribeiro S, Vrettou C, Koehler U, Griesinger G, Goossens V, Magli C, Albanese C, Parriego M, Coll L, Ron-El R, Sermon K, Traeger-Synodinos J. Aneuploidy in oocytes from women of advanced maternal age: analysis of the causal meiotic errors and impact on embryo development. Hum Reprod. 2023 Dec 4;38(12):2526-2535. doi: 10.1093/humrep/dead201. PMID 37814912
- [Derived] Verpoest W, Staessen C, Bossuyt PM, Goossens V, Altarescu G, Bonduelle M, Devesa M, Eldar-Geva T, Gianaroli L, Griesinger G, Kakourou G, Kokkali G, Liebenthron J, Magli MC, Parriego M, Schmutzler AG, Tobler M, van der Ven K, Geraedts J, Sermon K. Preimplantation genetic testing for aneuploidy by microarray analysis of polar bodies in advanced maternal age: a randomized clinical trial. Hum Reprod. 2018 Sep 1;33(9):1767-1776. doi: 10.1093/humrep/dey262. PMID 30085138